CLINICAL TRIAL: NCT04463212
Title: Systemic Endothelial Dysfunction in Reversible Cerebral Vasoconstriction Syndrome : a Case Control Study
Brief Title: Endothelial Dysfunction in Reversible Cerebral Vasoconstriction Syndrome
Acronym: DESS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0280
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Reversible Cerebral Vasoconstriction Syndrome
Keywords: Endothelial dysfunction; Reversible cerebral vasoconstriction syndrome; Arterial stiffness; Breath holding index; Pulse wave velocity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Diagnosis of probable SVCR evoked, faced with a single or repeated episode of unusual thunderclap or rapidly progressive headache, and demonstration of diffuse vasospasms via sectional imaging (angiography, angio-MRI or cerebral arteriography) or an increase in transcranial doppler speeds
- Subject control: Subject without SVCR (current and history)

SUMMARY:
Reversible Cerebral Vasoconstriction Syndrome (RCVS) is a syndrome described at the end of the 20th century. Generally, it has a benign course. It is revealed by acute headaches, in different circumstances such as sexual activity, physical exertion or emotional disturbances. But, in few cases, it might be complicated by seizure, stroke and subarachnoid haemorrhage. The diagnosis is confirmed on radiological examination, which shows diffuse cerebral vasoconstriction of brain vessel. It calls reversible because at three month, vasoconstriction disappears. Most cases occur during post partum or after serotoninergic/adrenergic drug use. The pathophysiology is unknown but a transient disturbance in the control of cerebrovascular tone by sympathic hyperactivity and/or endothelial dysfunction are suspected. The assessment of endothelial dysfunction in brain is possible with transcranial doppler. Chen et al. showed an impairment of vasodilatation post apnea induced called BHI on RCVS subjects compared with healthy control. BHI is a reflect of endothelial function in brain. Currently, investigators do not know if endothelial dysfunction occurred only in brain or if it may occur in systemic vessel. Some case reports talk about systemic complication such as kidney infarct or hepatic arterial vasospasm so a systemic vascular dysfunction may be suspected. In this study, researchers will study systemic endothelial function by measure of the pulse wave velocity during RCVS and after its recovering at 3 months, and compare it at healthy controls.

DETAILED DESCRIPTION:
The investigators lead a case control study to find a systemic endothelial dysfunction by the using of Complior device. Complior is a mechanographer who calculates pulse wave velocity (PWV). Pulse wave velocity is a reflect of arterial stiffness and it's correlate with endothelial dysfunction. For BHI, a Philips echograph is used before and after 30 second of breath holding.

Study protocol is :

For Patient :

* Day 0 : in hospital : anamnesis, medical history, physic examination, EKG, blood sample analysis, BHI, PWV analysis
* Month 1 : in medical visit : medical evolution, physic examination, EKG, blood sample analysis, BHI, PWV analysis
* Month 3 : in medical visit : medical evolution, physic examination, EKG, blood sample analysis, BHI, PWV analysis, cerebral angioCT Scan

For control :

- Day 0 : in hospital : medical history, physic examination, EKG, BHI, PWV analysis

ELIGIBILITY:
Inclusion Criteria for patients :

* Aged from 18 to 80 years old
* RVCS diagnosis evoked on clinic and radiologic finding
* Last headache was 15 days ago
* Oral consent
* Register in French social security

Inclusion criteria for control :

* Aged from 18 to 80 years old
* Hypothesis of RCVS in clinical presentation and on cerebral imaging
* Last headache less than 3 days old
* Oral consent
* Register in French social security
* Person under guardianship, curatorship or safeguarding of justice

Exclusion Criteria:

Non inclusion criteria for patient :

* Pregnant women
* Tobacco, coffee, alcohol, drugs or vasoactive recreational substances use within 2 hours prior to the examination.
* Person under guardianship, curatorship or safeguarding of justice
* Non sinusal rhythm on EKG
* Impossible of Breath holding for 30 secondes

Exclusion criteria for patient :

- No reversibility at 3 months

Non inclusion criteria for control :

* Pregnant women
* Tobacco, coffee, alcohol, drugs or vasoactive recreational substances use within 2 hours prior to the examination.
* Non sinusal rhythm on EKG
* Impossible of Breath holding for 30 secondes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Compare systemic endothelial function between patient and healthy subject | 24 hours
  By using Complior, researchers assess systemic endothelial function at inclusion on patient and healthy volunteer person by pulse wave velocity (cm.s-1)

SECONDARY OUTCOMES:
BHI (Breath Holding Index) | at day 0, month 1, month 3
  BHI measure on middle cerebral arteries by transcranial ultrasound
Pulse wave velocity (PWV) | at day 0, month 1, month 3
  Pulse wave velocity mesaure from carotid to femoral artery
Relationship between cerebral and systemic endothelial function | at day 0, month 1, month 3
  Comparison of BHI and VOP evolution
Renal failure | Day 0
  Diminution of creatinin clearance<100 ml/min/1.73m2
Occurence of stroke or cerebral oedema | at day 0, month 1, month 3
  Occurrence of ischemic stroke, cerebral haemorrhage, cerebral oedema
Comparison of PWV between patients with or without arterial hypertension | at day 0, month 1, month 3
  Comparison between middle PWV (cm/s) of patients with arterial hypertension and patients without arterial hypertension
Comparison of BHI between patients with or without arterial hypertension | at day 0, month 1, month 3
  Comparison between middle BHI of patients with arterial hypertension and patients without arterial hypertension
Comparison between PWV (cm/s) | at 3 months
  Comparison between PWV (cm/s) between patients and control group
Comparison between BHI (cm/s) | at 3 months
  Comparison between BHI (cm/s) between patients and control group

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Constant Dit Beaufils P, Barbin L, Pere M, Colleu C, Connault J, Preterre C, Guillon B, de Gaalon S. Systemic Arterial Stiffness in Reversible Cerebral Vasoconstriction Syndrome: A Prospective Case-Control Study. Eur J Neurol. 2026 Feb;33(2):e70495. doi: 10.1111/ene.70495. PMID 41589411